CLINICAL TRIAL: NCT04400773
Title: The Impact of Upper Body Plyometrics on Junior Male Cricket Fast Bowlers' Delivery Speed in Guyana
Brief Title: Upper Body Plyometrics in Junior Male Cricket Fast Bowlers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Sharmella Roopchand-Martin, Head- Mona Academy of Sport, The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ECP19-18-19
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Sport Performance
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: Two group pre-test post-test.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric Group (Experimental): This group will receive a 6-week upper body plyometric exercise protocol. Sessions will last for 65 minutes, three times per week. Each week the exercises will be progressed and all sessions will be supervised by an exercise professional.
  Interventions: Other: Plyometric exercises
- Strength Group (Experimental): This group will receive a 6-week upper body strength exercise protocol. Sessions will last for 65 minutes, three times per week. Each week the exercises will be progressed and all sessions will be supervised by an exercise professional.
  Interventions: Other: Strength training exercises

INTERVENTIONS:
Other: Plyometric exercises — Types of exercises include resistance tubing 90-90 external rotation, plyometric push-up, reverse overhead throws, rotational wall throw, overhead medicine ball, chest passes.
  Arms: Plyometric Group
Other: Strength training exercises — Types of exercise include push-ups, resisted external rotation, overhead presses, biceps curl, bench presses and triceps kick backs.
  Arms: Strength Group

SUMMARY:
A six-week upper body plyometric training program will be used to investigate its impact on fast bowling speed in junior male cricket players in Guyana, using a Stalker Sport 2 radar gun.

DETAILED DESCRIPTION:
This randomized pilot study will compare the effects of a six-week Upper Body Plyometric program with Upper Body Strength Training. After gaining ethical approval and baseline bowling speeds recorded, thirty under 19 club level fast bowlers will be assigned to two groups to complete either an upper-body plyometric or strength training program. Each group will participate in three (3) supervised exercise intervention sessions per week. Each 65-minute session will consist of a warm-up and cool-down program in addition to specific and routinely progressed upper body exercises as per each group's protocol. At the end of the intervention period, their bowling speeds will again be measured using a Stalker Sport 2 radar gun.

ELIGIBILITY:
Inclusion Criteria:• Only male athletes were admitted to the study.

* Athletes must have been practicing the art of fast bowling for at least one year at the club level.
* Athletes must have been between the ages of 15-19.
* Athletes must have been uninjured at the time of commencement of the study.

Exclusion Criteria:

* • Were outside of the age group being surveyed at the time of the study,

  * Had been practicing fast bowling at the club level for less than one (1) year,
  * Was injured at the time of commencement or within one year of the study.
  * Could not commit to full participation in the study's training regimes.
  * Received surgery in the three years prior to the study or had undergone rehabilitation within the past year.
  * Were currently engaged in plyometric training as this may confound the study.

Ages: 15 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Bowling speed | After 6 weeks of exercise training
  Cricket fast bowlers' bowling speed measured using the Stalker Sport 2 radar gun

CONTACTS AND LOCATIONS:
Locations (1):
- Cricket Association-Clubs, Georgetown, Guyana

IPD SHARING:
Plan to Share IPD: No